CLINICAL TRIAL: NCT01115361
Title: Improving Access to and Uptake of Postpartum Family Planning Service Through Enhanced Family Planning in Immunization Services
Brief Title: Postpartum Family Planning Service Through Enhanced Family Planning in Immunization Services
Acronym: PPFP-IZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Ministry of Health, Rwanda (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 890028
Record Dates: First submitted 2010-04-28; First posted 2010-05-04 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Contraception
Keywords: family planning; postpartum; immunization; integration; Contraceptive behavior
MeSH Terms: conditions — Contraception Behavior | interventions — Family Planning Services; Postpartum Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPFP in child immunization (Experimental): Women attending immunization services for their infant will receive educational brochures, group education and individual counseling on the benefits of the health timing and spacing of births,, pregnancy risk and return to fertility during the extended postpartum period (12 months), and referral to family planning services for those who are interested.
  Interventions: Behavioral: Family planning for postpartum women
- Control - Standard of care (No Intervention): The control arm will receive standard of care infant immunization services.

INTERVENTIONS:
Behavioral: Family planning for postpartum women — A.Group education sessions regarding pregnancy risk, benefits of FP, and family planning options during the postpartum period.
  B. IEC materials that deliver messages about the benefits of spacing pregnancies by at least 2 years, LAM, return to fecundity and pregnancy risk during the postpartum period and contraceptive options for postpartum women.
  C. Use of a screening tool to assess pregnancy risk for postpartum women coupled with a brief counseling message and referral to FP services.
  D.Convenient offer of FP services to women attending vaccination services for their infants.
  Arms: PPFP in child immunization

SUMMARY:
The purpose of this study is to determine the effectiveness of an intervention, which is designed to increase contraceptive prevalence among postpartum women attending vaccination services who desire to either space or limit their pregnancies, thus reducing unmet contraceptive need in this population.

DETAILED DESCRIPTION:
Study Goal:

To determine the effectiveness of an intervention, which is designed to increase contraceptive prevalence among postpartum women attending vaccination services who desire to either space or limit their pregnancies, thus reducing unmet contraceptive need in this population.

The Intervention:

A. Brief, concise messages conveyed to women during group education sessions regarding pregnancy risk, benefits of FP, and family planning options during the postpartum period.

B.IEC materials such as posters and brochures that deliver messages about the benefits of spacing pregnancies by at least 2 years, LAM, return to fecundity and pregnancy risk during the postpartum period and contraceptive options for postpartum women.

C.Use of a screening tool (Appendix A) to assess pregnancy risk for postpartum women coupled with a brief counseling message depending upon risk classification which includes referral to FP services for those currently or soon-to-be at-risk of pregnancy.

D.Convenient offer of FP services to women attending vaccination services for their infants either concurrently with vaccination services, or at the same facility and on the same day, but at a different time from vaccination services.

Study Design:

Experimental, two-group (intervention/control) pretest (pre-intervention) /posttest (post-intervention) design 12 month intervention period. A mid-course collection of process data will also be conducted at 6 months to assess the degree to which the intervention is being implemented as intended and to provide an opportunity for corrective action if needed.

Participants: Women attending vaccination services for their infants, and vaccination and FP providers

ELIGIBILITY:
Inclusion Criteria:

Clients:

* adult women, aged 21 years and older, or married women ages 18 to 20 who have achieved legal majority status by emancipation due to marriage,
* bring their infants between the ages 6-12 months to immunization services at study sites

Providers:

* all health care providers who currently provide immunization services to infants and/or family planning services within the selected facilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Use of a modern contraceptive method among postpartum women | 1 year
  The outcome variable is a dichotomous variable - use of modern FP method: yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S Dulli, PhD, MHS, Principal Investigator — FHI 360; Steve Sortijas, MPH, Study Director — FHI 360; Fidèle Ngabo, MD, MPH, Principal Investigator — Ministry of Health, Rwanda
Locations (1):
- Rwanda health care facilities, Kigali, Rwanda